CLINICAL TRIAL: NCT05772247
Title: Predictive Value of PS Application in Premature Infants With RDS by Different Pulmonary Ultrasound Scores: a Prospective Multicenter Study
Brief Title: Predictive Value of PS Application in Premature Infants With RDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: FirstJilinU2
Record Dates: First submitted 2023-02-12; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PS application
  Interventions: Diagnostic Test: Lung ultrasound
- non-PS application
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound score was calculated by the results of lung ultrasound examination

SUMMARY:
A multicenter prospective study was conducted to compare the predictive value of 6-zone, 10-zone, and 12-zone LUS scores for PS application in early and late preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission within 2 hours after birth;
2. The diagnosis was RDS;
3. Parents agree to attend

Exclusion Criteria:

1. chromosomal abnormalities or complex congenital malformations;
2. congenital pulmonary disease;
3. severe sepsis, disseminated intravascular coagulation, septic shock and other critical conditions;
4. LUS and blood gas analysis have been examined before the application of alveolar surfactant.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants <37 weeks gestational age
Sampling Method: Non-Probability Sample
Enrollment: 1392 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether the patient uses ps (pulmonary surfactant) | 2023.2-2023.12
  The standards used by PS are based on the European consensus